CLINICAL TRIAL: NCT05372783
Title: A Randomized, Placebo-Controlled Trial to Evaluate the Efficacy of Intranasal STI-9199 in Treating Symptomatic COVID-19 in Outpatient Adults and Adolescents
Brief Title: Study to Evaluate the Efficacy of IN STI-9199 in Treating Symptomatic COVID-19 in Outpatient Adults and Adolescents
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was never launched
Sponsor: Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHLD-COV-201
Record Dates: First submitted 2022-05-10; First posted 2022-05-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: COVID-19
Keywords: covid-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- STI-9199 (Experimental): 4 mg, 10 mg or 20 mg STI-9199 administered intranasally
  Interventions: Drug: STI-9199
- Placebo (Placebo Comparator): Placebo administered intranasally
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: STI-9199 — STI-9199 is a fully human monoclonal antibody which is a neutralizing antibody to SARS-CoV-2
  Arms: STI-9199
Drug: Placebo — Diluent solution
  Arms: Placebo

SUMMARY:
This is a Phase 2 global, randomized, double-blind, placebo-controlled study designed to investigate the safety and preliminary efficacy of intranasal STI-9199 in adults and adolescents who are COVID-19 positive with mild to moderate symptoms.

DETAILED DESCRIPTION:
This is a Phase 2 global, randomized, double-blind, placebo-controlled study designed to investigate the safety and preliminary efficacy of intranasal STI-9199 in adults and adolescents who are COVID-19 positive with mild to moderate symptoms. This is a single dose study and three different dose concentrations will be compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy, positive for COVID-19 by an EUA-approved rapid antigen or PCR test, has ongoing "mild to moderate illness or symptoms" with symptom onset starting < 5 days prior to screening visits
* Must provide written informed consent/assent if a minor which includes signing the institutional review board/independent ethics committee approved consent form prior to participating in any study related activity
* Willing and able to comply with study procedures and follow-up visits
* Willing to follow all contraception guidelines

Exclusion Criteria:

* In the Investigator's opinion, has progressive symptoms with likely imminent (24-48 hours) hospitalization or severe COVID-19 illness/symptoms
* Any medical condition that, in the Investigator's or designee's opinion, could adversely impact participant safety or key objectives of the study
* Has a prior history of long COVID
* Has a clinically documents acute infection other than COVID-19
* Known or suspected pregnancy, planned pregnancy, a positive pregnancy test at screening or are breastfeeding
* Has participated, or is participating in a clinical reserach study evaluating COVID-19 convalescent plasma, mAbs against SARS-CoV-2, or IV immunoglobulin within 2 months or less than 5 half-lives of the investigational product (whichever is longer) prior to the screening visit

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Change in viral load | Baseline through Day 8
  Change in viral load from baseline to Day 8 based on quantitative reverse-transcription polymerase chain reaction of COVID-19 virus from oropharyngeal swab collection
Incidence of adverse events (AEs) (safety) | Baseline through study completion at up to 30 days
  Safety as assessed by incidence of AEs by type, frequency, severity, and causality using the FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials

SECONDARY OUTCOMES:
Change in viral load | Baseline through Day 11
  Change in viral load from baseline to Day 4, Day 11 and Day 15 based on quantitative reverse-transcription polymerase chain reaction of COVID-19 virus from oropharyngeal swab collection
Participant perceived disease progression | Baseline through Day 15
  Participants rate their progression of disease on Day 8 and Day 15 when asked "Have your COVID symptoms gotten worse since treatment?" Yes or No response
Rate of COVID-19-related medical visits | Baseline through Day 30
  Determine the proportion of participants having COVID-19-related medically attended visits, emergency department assessments, hospitalization or all-cause mortality
Patient rated response | Baseline through D15
  Proportion of participants scoring ≥ +1 and those scoring ≤ -1 using a patient global impression of change (PGIC) 7-point categorical scale on Day 8 and Day 15 when responding to the question "In terms of your COVID-19 symptoms, how much benefit if any did you receive from the treatment?" The 7-point scale range is -3 to +3 where -3 is "very much worse" to +3 "very much improved" based on how the participant feels post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mike Royal, MD, Study Director — Sorrento Therapeutics, Inc.
Locations (1):
- ProSciento, Inc., Chula Vista, California, United States